CLINICAL TRIAL: NCT05439746
Title: Clinical Trial to Assess the Efficacy of Microlyte Matrix on the Healing of Surgically Created Partial Thickness Donor Site Wounds on Patients Requiring Split-thickness Skin Grafting
Brief Title: A Study to Evaluate the Efficacy of Microlyte Matrix in the Management of Donor Site Wounds
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Imbed Biosciences (Industry)
Collaborators: Arizona Burn Center, Maricopa Medical Center (Phoenix, AZ) (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Imbed 01
Record Dates: First submitted 2022-06-01; First posted 2022-06-30 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Wounds and Injuries
Keywords: Donor; Skin Graft; Wound; Partial Thickness
MeSH Terms: conditions — Wounds and Injuries

STUDY DESIGN:
Masking Description: The primary outcome assessment in this trial will be assessed by digital photography of the wounds as assessed by study team members who are blinded to the randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Matrix Comparison (Experimental): Qualified subjects are randomly assigned Microlyte Matrix in an open label fashion to half of a randomized similar depth donor site areas within a subject and determining percent healing at Day 14.
  Interventions: Device: Microlyte® Matrix

INTERVENTIONS:
Device: Microlyte® Matrix — Microlyte® Matrix is indicated for the management of wounds and can be used over-the-counter for minor wounds such as abrasions and lacerations, minor cuts, and minor scalds and burns. Under the direction of a healthcare professional, Microlyte® Matrix may be used for more serious wounds such as partial and full thickness pressure ulcers, venous stasis ulcers, diabetic ulcers, first and second-degree burns, abrasions and lacerations, donor sites and surgical wounds. Microlyte® Matrix may be used over debrided and grafted partial thickness wounds.

SUMMARY:
A study to to evaluate the efficacy of Microlyte® Matrix by demonstrating its superiority to the standard of care in the healing of donor site wounds in patients requiring split-thickness grafting, as well as to assess the occurrence of donor site wound infection, allergic reaction, pain and itching, and scarring at 12 weeks, assessed by patients using the Patient and Observer Scar Assessment Scale (POSAS).

DETAILED DESCRIPTION:
The proposed study is a randomized, controlled, open-label clinical trial to assess the efficacy in wound healing of the FDA 510k cleared Microlyte® Matrix (K153756) in surgically created partial thickness donor site wounds > 100 cm2 in size on patients and harvested at 12/1000th inch requiring split-thickness skin grafting. Subjects are expected to be hospitalized as in-patients for approximately 7 days following initial donor site surgery. Study visits conducted after hospital discharge must be conducted as out-patient clinic visits.

Each wound will be divided into proximal and distal halves with one half randomized to receive Microlyte® Matrix. Kaltostat/Tegaderm will be used as the control. Thus, each patient is their own control removing the potential variability of the depth of donor site wounds between patients as a confounding factor.

Microlyte® Matrix is a FDA-cleared (K153756) antimicrobial dressing manufactured by Imbed Biosciences, Inc. (Madison, WI), which is an ISO 13485 certified/FDA QSR compliant facility. It is indicated for the management of partial and full thickness wounds including pressure ulcers, venous stasis ulcers, diabetic foot ulcers, first and second-degree burns, abrasions and lacerations, donor sites and surgical wounds.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients where creation of a donor site wound for any indication including chronic wound, burn wound, surgical/traumatic wound, and tumor excision.
2. Donor site wound with a surface area of greater than 100 cm2 is required.
3. At least 18 years of age
4. Provision of signed and dated informed consent form
5. Stated willingness to comply with all study procedures and availability for the duration of the study
6. Ability and willingness to adhere to the study intervention regimen and follow-up visits

Exclusion Criteria:

1. Age less than 18 years.
2. Vulnerable population.
3. Pregnant, lactating or nursing women.
4. Unable to provide consent.
5. Presumed unable to complete follow-up assessments.
6. Prior adverse reaction or sensitivity to silver.
7. Enrollment in another interventional trial using a systemic therapeutic within 30 days prior to enrollment for this study.
8. Presumed impairment of wound healing as with prescription drugs or medical diagnoses that have potential to impair wound healing at the discretion of clinical investigator, e.g., cancer, transplant status, autoimmune disease, severe malnutrition, etc.
9. Any diagnosis with concern for 30 Day mortality.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 53 (Estimated)
Dates: Start 2023-01-01 (Estimated); Primary Completion 2024-01-30 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of donor site wound closure | Day 14 post-op
  Therefore, assessment of the percentage wound closure at the time of primary outcome assessment (14 days) provides a very reliable method for detection of differences between groups. Digital photography and Image-J analysis allow for blinded assessment of primary outcome.

SECONDARY OUTCOMES:
Percentage of donor site wound closure | Day 7 post-op
  Signs of infection or allergic reactions, pain, and pruritus assessed during each study visit.
Durability of wound closure, assessed by percentage of wound closure | 12 weeks
  Wound Closure ranges from 0%-100% with 0% being no wound closure occurring and 100% being full closure
Pain, itching, and scarring, assessed by patients using the Patient and Observer Scar Assessment Scale (POSAS). | 12 weeks
  POSAS Scale is a series of questions with answers ranging from 1-10, with 1 dictating few or negligible differences from normal skin, and 10 being unimaginable scar difference from normal skin.
Signs of infection or allergic reactions, pain, and pruritus | 12 weeks

IPD SHARING:
Plan to Share IPD: No